CLINICAL TRIAL: NCT02000180
Title: Do Progressive Levels of Simulation Fidelity Enhance Colonoscopic Skill Acquisition and Transfer in Novice Endoscopic Trainees?
Brief Title: Colonoscopic Skill Acquisition and Transfer Via Simulated Curriculum of Progressive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Samir Grover, Staff Physician/Assistant Professor, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 13-060
Record Dates: First submitted 2013-11-17; First posted 2013-12-04 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Group (Experimental): The progressive learning group will undertake 6 hours of interactive small-group didactic sessions, interlaced with up to 6 hours of self-directed instruction initially on the low-fidelity box simulator, with feedback provided one-on-one by an expert academic endoscopist. Participants in the progressive learning group can switch to the high-fidelity simulator at their discretion, but cannot return to the low-fidelity simulator. On the high fidelity VR simulator they can progress through six modules each in colonoscopy and endoscopic polypectomy in a self-directed fashion, with one-on-one feedback by an expert academic endoscopist. The endoscopy instructor will demonstrate techniques, answer questions and provide feedback. The entirety of this will be delivered over two days.
  Interventions: Behavioral: Progressive Group
- High-Fidelity Group (No Intervention): The high-fidelity group will undertake 6 hours of interactive small-group didactic and hands-on sessions on the theory of colonoscopy, led by an expert academic gastroenterologist. The sessions will be interlaced with up to six hours of self-directed instruction on the high-fidelity VR simulator. Six task-specific modules of increasing difficulty in colonoscopy and colonoscopic polypectomy will be taught solely on the VR simulator with one-on-one feedback from an expert academic endoscopist. The endoscopy instructor will demonstrate techniques, answer questions and provide feedback as necessary. The entirety of this will be delivered over two days.

INTERVENTIONS:
Behavioral: Progressive Group
  Arms: Progressive Group

SUMMARY:
It is hypothesized that a progressive simulated learning strategy will result in better global clinical performance (e.g., technical, communication) and transfer of endoscopic skill, as compared with a high-fidelity simulation strategy.

ELIGIBILITY:
Inclusion Criteria:

* novice endoscopists from Adult Gastroenterology, Pediatric Gastroenterology, General Surgery training programs at University of Toronto

Exclusion Criteria:

* Trainees who have performed greater than 25 colonoscopies will be excluded to ensure all participants are novices.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir C Grover, MD/MEd, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grover SC, Scaffidi MA, Khan R, Garg A, Al-Mazroui A, Alomani T, Yu JJ, Plener IS, Al-Awamy M, Yong EL, Cino M, Ravindran NC, Zasowski M, Grantcharov TP, Walsh CM. Progressive learning in endoscopy simulation training improves clinical performance: a blinded randomized trial. Gastrointest Endosc. 2017 Nov;86(5):881-889. doi: 10.1016/j.gie.2017.03.1529. Epub 2017 Mar 31. PMID 28366440

RESULTS

PARTICIPANT FLOW:
Groups:
- Progressive Group: The progressive learning group will undertake 6 hours of interactive small-group didactic sessions, interlaced with up to 6 hours of self-directed instruction initially on the low-fidelity box simulator, with feedback provided one-on-one by an expert academic endoscopist. Participants in the progressive learning group can switch to the high-fidelity simulator at their discretion, but cannot return to the low-fidelity simulator. On the high fidelity VR simulator they can progress through six modules each in colonoscopy and endoscopic polypectomy in a self-directed fashion, with one-on-one feedback by an expert academic endoscopist. The endoscopy instructor will demonstrate techniques, answer questions and provide feedback. The entirety of this will be delivered over two days.
  Progressive Group
Period: Overall Study
Arm/Group | Progressive Group | High-Fidelity Group
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progressive Group | High-Fidelity Group | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (3) | 28.1 (2) | 28.1 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 13 | 10 | 23
Training program (gastroenterology, general surgery, or internal medicine) [Count of Participants; unit: Participants]
  Gastroenterology | 6 | 4 | 10
  General surgery | 11 | 14 | 25
  Internal medicine | 1 | 1 | 2
Endoscopic experience [Mean (Standard Deviation); unit: Number of procedures]
  Independent colonoscopies completed before trainin | 0.8 (2.8) | 0.2 (0.8) | 0.5 (1.8)
  Assisted colonoscopies completed before training | 5.5 (13.7) | 3.6 (3.4) | 4.5 (8.5)
  Indendent EGDs completed before training | 1.8 (5.5) | 0.9 (1.7) | 1.3 (3.6)
  Assisted EGDs completed before training | 6 (13.5) | 3.2 (4.6) | 4.6 (9.0)
  Independent colonoscopies completed after training | 0.1 (0.3) | 0 (0) | 0.1 (0.1)
  Assisted colonoscopies completed after training | 1.5 (1.9) | 2 (3.6) | 1.7 (2.7)
  Independent EGDs completed after training | 0.4 (1) | 0.2 (0.7) | 0.3 (0.8)
  Assisted EGDs completed after training | 1.3 (2.3) | 2 (3.5) | 1.7 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Progressive and High-Fidelity Groups on Clinical Colonoscopy Peformance (JAG/DOPS)
Description: The Joint Advisory Group (JAG) Direct Observation of Procedural Skills (DOPS) tool is a tool to assess colonoscopic competency and includes ratings of the following domains: (i) assessment, consent and communication; (ii) safety and sedation; (iii) endoscopic skills during insertion and withdrawal; and, (iv) diagnostic and therapeutic ability. Scores range from 0-100, with higher scores representing higher colonoscopic competency. The tool will be used to assess participants before and after the intervention at a time of one week. A change in these ratings before and after intervention is the primary outcome.
Time Frame: 4-6 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progressive Group | High-Fidelity Group
Number analyzed (Participants) | 18 | 19
units on a scale
  Procedure 1 | 68.2 (6.9) | 59.0 (7.2)
  Procedure 2 | 68.3 (6.1) | 59.1 (8)

2. Secondary Outcome: Cognitive Knowledge of Endoscopy
Description: Assessed via a multiple-choice question test on the theory and practice of endoscopy. Scores range from 0-100 with higher scores representing a more knowledge of the theory and practice of endoscopy.
Time Frame: Pre-training, immediate post-training
Measure: Mean (Standard Deviation); unit: percentage score on MCQ test
Arm/Group | Progressive Group | High-Fidelity Group
Number analyzed (Participants) | 18 | 19
percentage score on MCQ test
  Pre-training | 36.2 (14.4) | 28.6 (12.6)
  Immediate post-training | 59.5 (6.8) | 59.5 (5.4)

3. Secondary Outcome: Colonoscopy Specific-performance.
Description: The Joint Advisory Group (JAG) Direct Observation of Procedural Skills (DOPS) tool is a tool to assess colonoscopic competency and includes ratings of the following domains: (i) assessment, consent and communication; (ii) safety and sedation; (iii) endoscopic skills during insertion and withdrawal; and, (iv) diagnostic and therapeutic ability. Scores range from 0-100, with higher scores representing higher colonoscopic competency. The tool will be used to assess participants on virtual reality colonoscopy cases. A change in these ratings before and after intervention is a secondary outcome.
Time Frame: Pre-training, immediate post-training, and 4-6 weeks after training (delayed post-training)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progressive Group | High-Fidelity Group
Number analyzed (Participants) | 18 | 19
units on a scale
  Pre-training | 22.04 (21.18) | 21.05 (22.61)
  Immediate post-training | 75.74 (16.99) | 65.96 (13.90)
  Delayed post-training | 90.74 (12.71) | 77.54 (16.92)

4. Secondary Outcome: Colonoscopy Specific Performance, Communication Skills, and Global Performance on an Integrated Scenario
Description: Technical skills, communication skills, and global performance assessed during an integrated scenario through the JAG DOPS tool, integrated scenario communication rating form (ISCRF), and integrated scenario global rating form (ISGRF) respectively.
  The JAG DOPS tool, as previously described, will be used to assess participants on integrated scenario colonoscopy cases. A change in these ratings before and after intervention is a secondary outcome.
  The ISCRF and ISGRF are tools which measure communication skills and global performance with a standardized nurse and standardized patient during a simulated colonoscopy. These tools can have scores from 0-100, with higher scores representing better performance.
Time Frame: Immediate post-training and 4-6 weeks after training (delayed post-training)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progressive Group | High-Fidelity Group
Number analyzed (Participants) | 18 | 19
units on a scale
  Immediate post - Colonoscopy specific performance | 68.88 (18.68) | 56.69 (13.47)
  Immediate post - Communication skills | 73.89 (11.7) | 67.89 (14.27)
  Immediate post - Global performance | 73.15 (12.6) | 66.75 (8.94)
  Delayed post - Colonoscopy specific performance | 87.08 (11.77) | 75.20 (17.30)
  Delayed post - communication skills | 83.33 (11.25) | 69.21 (13.15)
  Delayed post - global performance | 80.13 (11.82) | 70.33 (9.60)

ADVERSE EVENTS:
Arm/Group | Progressive Group | High-Fidelity Group
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No